CLINICAL TRIAL: NCT04080453
Title: Pro-inflammatory Role of Blood Platelets in Critically Ill Patients With Septic Shock: an Observational Study.
Brief Title: Pro-inflammatory Role of Blood Platelets in Critically Ill Patients With Septic Shock.
Acronym: PLAQSIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: MSD France (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2017/20
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Septic Shock
Keywords: Blood platelets; CD40 ligand; Multiple Organ Failure
MeSH Terms: conditions — Shock, Septic; Hyper-IgM Immunodeficiency Syndrome; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic shock: Plasma of 100 patients presenting a septic shock will be analysed including plasma concentration in CD154, beta thromboglobulin, platelet factor 4, platelet microparticles, soluble CD62, RANTES, GRO-alpha and HMGB-1
  Interventions: Other: Septic shock
- Systemic Inflammatory Response Syndrome: Plasma of 100 patient presenting a systemic inflammatory response syndrome = SIRS will be analysed including plasma concentration in CD154, beta thromboglobulin, platelet factor 4, platelet microparticles, soluble CD62, RANTES, GRO-alpha and HMGB-1
  Interventions: Other: Systemic Inflammatory Response Syndrome

INTERVENTIONS:
Other: Septic shock — Plasma concentration in CD154, beta thromboglobulin, platelet factor 4, platelet microparticles, soluble CD62, RANTES, GRO-alpha, HMGB-1, monocyte Dnases signal, circulating free DNA and DNase1 and DNase1L3 activities will be studied and compared at inclusion (Day 0), Day 1 and Day 5.
  Groups: Septic shock
Other: Systemic Inflammatory Response Syndrome — Plasma concentration in CD154, beta thromboglobulin, platelet factor 4, platelet microparticles, soluble CD62, RANTES, GRO-alpha, HMGB-1, monocyte Dnases signal, circulating free DNA and DNase1 and DNase1L3 activities will be studied and compared at inclusion (Day 0), Day 1 and Day 5.
  Groups: Systemic Inflammatory Response Syndrome

SUMMARY:
Blood platelets play a major role in the inflammatory response. A dysregulation of platelets activation may be one of the contributors to tissue damage in critically ill patients with septic shock. The main objective of this study is to compare platelet activation markers levels (including plasma concentration in CD154, beta thromboglobulin, platelet factor 4, platelet microparticles, soluble CD62, RANTES, GRO-alpha and HMGB-1) at the early phase of a septic shock and a systemic inflammatory response syndrome (SIRS).

DETAILED DESCRIPTION:
Sepsis is defined as life-threatening organ dysfunction due to dysregulated host response to infection which can lead to many failures of vital organs (kidneys, lungs, liver) in critically ill patients. It is accompanied at an early phase by both a proinflammatory and procoagulant state generating many platelet activators. Given their essential role in the inflammatory response, a dysregulation of platelets activation may be one of the contributors to tissue damage. To determine if platelet activation contribute to deregulation of the inflammatory response of the host in sepsis, the main objective of this study is to compare platelet activation markers levels of patients with septic shock and after major surgery. Plasma concentration in CD154, beta thromboglobulin, platelet factor 4, platelet microparticles, soluble CD62, RANTES, GRO-alpha, HMGB-1, monocyte Dnases signal, circulating free DNA and DNase1 and DNase1L3 activities will be studied and compared at inclusion (Day 0), Day 1 and Day 5.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years admitted to an intensive care unit for:

  * a septic shock evolving for less than 24h (defined by an increase in the SOFA (Sequential Organ Failure Assessment) score of at least 2 points related to an infection, a persisting hypotension requiring vasopressors to maintain MAP ≥65 mmHg and a serum lactate level >2 mmol/L (18 mg/dL) despite adequate volume resuscitation)
  * Or a systemic inflammatory response syndrome (SIRS) evolving for less than 24h (defined as 2 or more of the following variables: fever of more than 38°C or less than 36°C, heart rate of more than 90 beats per minute, respiratory rate of more than 20 breaths per minute or arterial carbon dioxide tension (PaCO2) of less than 32 mm Hg, abnormal white blood cell count (>12,000/µL or <4,000/µL or >10% immature forms).

Exclusion Criteria:

* Age < 18 years
* Known history of constitutional thrombopathy (Bernard Soulier's disease, Glanzmann thrombasthenia, Gray's syndrome or dense granule disease)
* Myeloproliferative or myelodysplastic syndrome
* Autoimmune thrombocytopenic purpura
* Acute leukemia
* Haemorrhagic shock
* Platelet transfusion within 7 days prior to inclusion
* Antiplatelet medication (clopidogrel or ticagrelor taken within 5 days of inclusion, prasugrel or dipyridamole within 7 days of inclusion)
* Active HIV infection or known active hepatitis B or C
* Pregnant or breastfeeding woman
* Patients protected by the law, under guardianship or trusteeship, or deprived of liberty
* Patients without health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, two populations will be recruiting, patients presenting a septic shock and patient presenting a SIRS, who will be admitted in intensive care unit or in continuing care units.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Plasma concentration | Day 0, day 1 and day 5
  Plasma concentration in CD154, beta thromboglobulin, platelet factor 4, platelet microparticles, soluble CD62, RANTES, GRO-alpha and HMGB-1 will be measured in each group by dosage

SECONDARY OUTCOMES:
Neutrophil Extracellular Traps formation | Day 0, day 1 and day 5
  Monocyte Dnases signal, circulating free DNA and DNase1 and DNase1L3 activities will be measured in each group by dosage
Markers of platelet activation and severity of organ failure | Day 0 and Day 7
  Correlation between markers of platelet activation and severity of organ failure will be measured by Sequential Organ Failure Assessment (SOFA) score.
  The score varies from 0 to 4.
Markers of platelet activation and inflammatory markers | Day 0 and Day 7
  Correlation between markers of platelet activation and inflammatory markers (leukocytes and CRP) will be measured by KDIGO score.The score varies from 1 to 4.
Markers of platelet activation and ISTH score | Day 0
  Correlation between markers of platelet activation and ISTH score of the International Society of Thrombosis and Haemostasis (ISTH) will be measured by Coagulation Intra Vasculaire Disséminée score. The score varies from < 5 to ≥ 5 :
  If score ≥ 5: compatible with a CIVD patent. If score <5: suggests a latent DIC.
Markers of platelet activation and platelet count | Day 0 and day 7
  Correlation between markers of platelet activation (CD154, beta thromboglobulin, platelet factor 4, platelet microparticles, soluble CD62, RANTES, GRO-alpha and HMGB-1) and platelet count.
Markers of platelet activation on ICU mortality | Day 0 and Day 7
  Prognostic aspect of markers of platelet activation (CD154, beta thromboglobulin, platelet factor 4, platelet microparticles, soluble CD62, RANTES, GRO-alpha and HMGB-1) on ICU mortality, hospital mortality, ICU and hospital length of stay, norepinephrine, kidney failure and ventilation free days.
Levels of platelet activation markers | Day 0 and Day 7
  Correlation between levels of platelet activation markers studied (CD154, beta thromboglobulin, platelet factor 4, platelet microparticles, soluble CD62, RANTES, GRO-alpha and HMGB-1).

CONTACTS AND LOCATIONS:
Overall Officials: Antoine DEWITTE, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Hôpital Haut Lévêque, Pessac, France